CLINICAL TRIAL: NCT06489730
Title: HAPH Registry: Time Course and Prognostic Significance of Pulmonary Artery Pressure in Highlanders.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Other Study IDs: HAPH_Register
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: High Altitude Pulmonary Hypertension; Sleep Apnea
Keywords: high altitude illness; pulmonary hypertension; sleep apnea; disease progression; hypoxia
MeSH Terms: conditions — Pulmonary edema of mountaineers; Sleep Apnea Syndromes; Hypertension, Pulmonary; Disease Progression; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Highlanders living above 2500 m: Highlanders permanently living above 2500 m in the Aksay area in Kyrgyzstan
- Low altitude control: Healthy lowlanders living below 1000 m.

SUMMARY:
The purpose of the current study is to evaluate the clinical and physiologic course of Kyrgyz highlanders with high altitude pulmonary hypertension (HAPH) by performing a longitudinal cohort study. To this end, the investigators will invite the same highlanders who participate din the study in 2017 to undergo follow-up examinations in 2024, in order to allow comparisons of current results with baseline data from 2017.

ELIGIBILITY:
Inclusion Criteria:

* Permanently living >2500 m
* Written informed consent

Exclusion Criteria:

* Highlanders who cannot follow the study investigations,
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, heavy smoking >20 cigarettes/day or >20 pack-years.
* Coexistent unstable systemic hypertension or coronary artery disease that required adjustment of medication within the last 2 months
* Regular use of medication that affects control of breathing (benzodiazepines, opioids, acetazolamide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Highlanders living at Aksay plateau will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary artery pressure in highlanders | Year 2017 to 2024
  Change in pulmonary artery pressure (RV/RA measured by echocardiography) from 2017 to 2024 in highlanders living above 2500 m.

SECONDARY OUTCOMES:
Change in pulmonary artery pressure between highlanders and lowlanders | Year 2017 to 2024
  Difference in the change in pulmonary artery pressure (RV/RA measured by echocardiography) from 2017 to 2024 between highlanders and lowland controls.
Change in TRP/CO in highlanders | Year 2017 to 2024
  Change in TRP/CO slope from 2017 to 2024 in highlanders living above 2500 m.
Progression of oxygen desaturation index | Year 2017 to 2024
  Change in the oxygen desaturation index from 2017 to 2024 in highlanders.
Progression of quality of life | Year 2017 to 2024
  Change in the mental and physical component score of the SF-36 questionnaire from 2017 to 2024 in highlanders.
Progression of arterial blood gases | Year 2017 to 2024
  Change in the arterial blood gases from 2017 to 2024 in highlanders.
Progression of right heart strain | Year 2017 to 2024
  Change in the right heart strain from 2017 to 2024 in highlanders.

CONTACTS AND LOCATIONS:
Overall Officials: Talant M Sooronbaev, Prof. Dr., Principal Investigator — National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov; Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology

IPD SHARING:
Plan to Share IPD: Undecided